CLINICAL TRIAL: NCT00002924
Title: Androgen Receptor Mutations in Hormone Refractory Prostate Cancer
Brief Title: Gene Mutations in Patients With Advanced Prostate Cancer That Is Not Responsive to Hormone Therapy
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-9663; U10CA031946 (NIH); CDR0000065329 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow biopsies were obtained from 164 patients enrolled on CALGB 9583 and from 20 patients enrolled on CALGB chemotherapy trials (CALGB 9480, 9680, 9780).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Source of patient samples: The CALGB conducted a phase III study (CALGB 9583) in which 260 men with AiPC were randomly assigned to antiandrogen withdrawal together with simultaneous ketoconazole and hydrocortisone versus antiandrogen withdrawal alone, followed by sequential ketoconazole and hydrocortisone. Metastatic disease with progression despite castrate levels of testosterone, prior antiandrogen therapy for a minimum of 4 weeks, and a minimum PSA level of 5 ng/mL were required; treatment with sequential antiandrogens was allowed. No prior chemotherapy was allowed. Bone marrow biopsies were obtained from 164 patients enrolled on CALGB 9583 and from 20 patients enrolled on CALGB chemotherapy trials (CALGB 9480, 9680, 9780).
  Interventions: Other: mutation analysis

INTERVENTIONS:
Other: mutation analysis

SUMMARY:
RATIONALE: Gene mutations may make prostate cancer cells unable to attach to androgens. This may permit the growth of prostate cancer. Gene testing may improve the identification of patients with advanced prostate cancer.

PURPOSE: Clinical trial to study the androgen receptor gene in patients with prostate cancer that is not responsive to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

1. the feasibility of collecting bone marrow biopsies from prostate cancer patients in a cooperative group setting
2. the incidence of marrow invasion by prostate tumor in random bone marrow biopsy
3. the influence of previous prostate radiation on obtaining prostate tumor
4. the frequency and type of AR mutations and
5. association of AR mutations with response to antiandrogen withdrawal.

ELIGIBILITY:
1. Histologically proven adenocarcinoma of the prostate that is refractory to hormone therapy
2. Patients who are eligible for anticancer therapy on Protocol CLB-9480, CLB-9583, CLB-9680, or CLB-9780 are also eligible for this study if they have not started treatment on those protocols

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible men enrolled on a trial of antiandrogen withdrawal had a minimum prostate-specific antigen (PSA) level of 5 ng/dL that was increasing on castration therapy including an antiandrogen. Marrow biopsies were obtained to collect prostate tumor. Additional samples were obtained from men enrolled on chemotherapy trials.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 1997-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 10 years

SECONDARY OUTCOMES:
response rate | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Study Chair — University of Massachusetts, Worcester
Locations (49):
- United States (49):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - St. Barnabas Medical Center, Livingston, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Ross RW, Halabi S, Ou SS, Rajeshkumar BR, Woda BA, Vogelzang NJ, Small EJ, Taplin ME, Kantoff PW; Cancer and Leukemia Group B. Predictors of prostate cancer tissue acquisition by an undirected core bone marrow biopsy in metastatic castration-resistant prostate cancer--a Cancer and Leukemia Group B study. Clin Cancer Res. 2005 Nov 15;11(22):8109-13. doi: 10.1158/1078-0432.CCR-05-1250. PMID 16299243
- [Result] Taplin ME, Rajeshkumar B, Halabi S, Werner CP, Woda BA, Picus J, Stadler W, Hayes DF, Kantoff PW, Vogelzang NJ, Small EJ; Cancer and Leukemia Group B Study 9663. Androgen receptor mutations in androgen-independent prostate cancer: Cancer and Leukemia Group B Study 9663. J Clin Oncol. 2003 Jul 15;21(14):2673-8. doi: 10.1200/JCO.2003.11.102. PMID 12860943
- [Result] Taplin ME, Halabi S, Rajeshkumar B, et al.: Androgen receptor mutations in androgen independent prostate cancer (APICA) do not correlate with anti-androgen withdrawal response: Cancer and Leukemia Group B (CALGB) 9663. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1738, 2001.
- [Result] Taplin ME, Rajeskumar B, Woda BA, et al.: Androgen receptor analyses in androgen independent prostate cancer (AIPCA): Cancer and Leukemia Group B (CALGB) 9663. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A1297, 2000.